CLINICAL TRIAL: NCT03939897
Title: A Randomized Phase I/II Trial of Fulvestrant and Abemaciclib in Combination With Copanlisib (FAC) Versus Fulvestrant and Abemaciclib Alone (FA) for Endocrine-Resistant, Hormone Receptor Positive, HER2 Negative Metastatic Breast Cancer (FAC vs FA)
Brief Title: Testing the Addition of Copanlisib to Usual Treatment (Fulvestrant and Abemaciclib) in Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-02752; NCI-2019-02752 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 201911082; 10287 (Other: Yale University Cancer Center LAO); 10287 (Other: CTEP); UM1CA186689 (NIH); UM1CA186704 (NIH)
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic HER2-Negative Breast Carcinoma; Metastatic Hormone Receptor-Positive Breast Carcinoma; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Biopsy; Specimen Handling; copanlisib; X-Rays; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I Part A Dose 1 (copanlisib, abemaciclib, fulvestrant) (Experimental): Patients receive 45 mg copanlisib hydrochloride IV over 1 hour on days 1 and 15 and 100 mg abemaciclib PO BID on days 2-28 of cycle 1 and on days 1-28 of subsequent cycles. Patients also receive 500 mg fulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Copanlisib Hydrochloride; Procedure: Diagnostic Imaging Testing; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Multigated Acquisition Scan
- Phase I Part A Dose 2 (copanlisib, abemaciclib, fulvestrant) (Experimental): Patients receive 45 mg copanlisib hydrochloride IV over 1 hour on days 1, 8, and 15 and 150 mg abemaciclib PO twice daily BID for 5 days each week (2 days off). Patients also receive f500 mg fulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Copanlisib Hydrochloride; Procedure: Diagnostic Imaging Testing; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Multigated Acquisition Scan
- Phase I Part B Dose 1b (copanlisib, abemaciclib, fulvestrant) (Experimental): Patients receive 45 mg copanlisib hydrochloride IV over 1 hour on days 1 and 15 and 100 mg abemaciclib PO twice daily BID for 5 days each week (2 days off). Patients also receive 500 fulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Copanlisib Hydrochloride; Procedure: Diagnostic Imaging Testing; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Multigated Acquisition Scan
- Phase I Part B Dose 2b (copanlisib, abemaciclib, fulvestrant) (Active Comparator): Patients receive 45 mg copanlisib hydrochloride IV over 1 hour on days 1, 8, and 15 and 100 mg abemaciclib PO twice daily BID for 5 days each week (2 days off). Patients also receive 500 mg fulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Copanlisib Hydrochloride; Procedure: Diagnostic Imaging Testing; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY 2835219; LY-2835219; LY2835219; Verzenio
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Copanlisib Hydrochloride — Given IV
  Other Names: 5-Pyrimidinecarboxamide, 2-Amino-N-(2,3-dihydro-7-methoxy-8-(3-(4-morpholinyl)propoxy)imidazo(1,2-C)quinazolin-5-yl)-, Hydrochloride (1:2); Aliqopa; BAY 80-6946 Dihydrochloride; BAY-80-6946 Dihydrochloride; Copanlisib Dihydrochloride
Procedure: Diagnostic Imaging Testing — Undergo imaging
  Other Names: Diagnostic Imaging; Medical Imaging
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ICI-182780; ICI182780; ZD 9238; ZD-9238; ZD9238
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning

SUMMARY:
This phase I trial studies the effects (good and bad) of adding copanlisib to the usual therapy of fulvestrant and abemaciclib in treating patients with hormone receptor positive and HER2 negative breast cancer that has spread from where it first started (breast) to other places in the body (metastatic). Some breast cancer cells have receptors for the hormones estrogen or progesterone. These cells are hormone receptor positive and they need estrogen or progesterone to grow. This can affect how the cancer is treated. Hormone therapy using fulvestrant may fight breast cancer by blocking the use of estrogen by the tumor cells. Abemaciclib and copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Adding copanlisib to the usual therapy of fulvestrant and abemaciclib may work better than giving fulvestrant and abemaciclib alone in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety profile of fulvestrant + abemaciclib + copanlisib hydrochloride (copanlisib) (FAC) and determine the recommended phase 2 dose (RP2D).

SECONDARY OBJECTIVES:

I. To assess the objective response rate (ORR = partial response [PR] + complete response [CR]) and clinical benefit rate (CBR = PR + CR + stable disease [SD] >= 6 months) of FAC and medium progression free survival (PFS) with FAC.

EXPLORATORY OBJECTIVES:

I. To assess whether triplet therapy with FAC inhibits AKT phosphorylation, reduces cyclin D1, and inhibits Rb phosphorylation.

II. To assess whether the combination of abemaciclib and fulvestrant affect the copanlisib pharmacokinetics (PK).

III. To assess the objective response rate (ORR), clinical benefit rate (CBR) and median PFS in the following molecularly defined subgroups treated with FAC such as mutations in genes in the PI3K pathway (PIK3CA, AKT, PTEN etc), ESR1, TP53, or PTEN IHC loss vs not.

IV. To assess baseline and treatment induced changes in various cancer associated pathways, including but not limited to PI3K, MAPK, ER, cyclins, CDKs and CDK inhibitors; and to correlate with treatment response and progression.

V. To correlate baseline and treatment induced changes in breast cancer intrinsic subtypes (PAM50), and PI3K messenger ribonucleic acid (mRNA) signature and expression of candidate genes with treatment response and benefit from adding copanlisib.

VI. To evaluate ctDNA mutations at baseline and over time for response predictors at baseline, and clonal evolution associated with treatment.

VII. To correlate ctDNA mutation profiles with tumor sequencing, and correlate baseline ctDNA mutations, particularly in components of the PI3K pathway with treatment response, and correlate early changes in ctDNA variant allele frequencies (VAFs) with PFS, assess emergent resistant mutations at progression.

VIII. To assess resistance mechanisms to FAC at baseline and at disease progression.

IX. To examine the molecular effects of FAC on tumor and circulating markers. X. To analyze tumor infiltrating lymphocytes at baseline, during treatment, and at disease progression.

OUTLINE: This is a phase I two part, dose-escalation study of copanlisib hydrochloride and abemaciclib.

PHASE I (PART A): Patients receive copanlisib hydrochloride intravenously (IV) over 1 hour on days 1, 8, and 15 or days 1 and 15 (depending on dose level) and abemaciclib orally (PO) twice daily (BID) on on days 2-28 of cycle 1 and on days 1-28 of subsequent cycles. Patients also receive fulvestrant intramuscularly (IM) on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an echocardiography (ECHO) or multigated acquisition (MUGA) scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.

PHASE I (PART B): Patients receive copanlisib hydrochloride IV over 1 hour on days 1, 8, and 15 or days 1 and 15 (depending on dose level) and abemaciclib PO twice daily BID for 5 days each week (2 days off). Patients also receive fulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.

After completion of study treatment, patients are followed up every 3 months for 5 years.

* As of November 2023, Bayer has decided to voluntarily withdraw the NDA for copanlisib, phase II portion removed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed ER and/or PR positive, HER2 negative or non-amplified breast cancer that is stage IV, with measurable or non-measurable disease. ER/PR positivity is defined as at least 1% positive or an Allred score of at least 3. HER2 status is defined per the 2018 American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guideline
* All patients must agree to provide archival tumor material for research and must agree to undergo research tumor biopsy before treatment if presence of easily accessible lesions (judged by the treating physician). For patients with bone only disease, or patients without easily accessible lesions for the baseline research biopsy, availability of archival tumor material (2 x 4-5 micron section unstained slides, plus 15-20 x 10 micron section unstained slides or a tumor rich block) from previous breast cancer diagnosis or treatment is required for central PTEN and PIK3CA analysis
* No more than 1 prior chemotherapy in the metastatic setting. There is no limit on prior lines of endocrine therapy. (For patients enrolling to the phase 1 portion of the study, prior fulvestrant, CDK4/6 inhibitor, and everolimus is allowed)
* For patients enrolling to the randomized phase 2 portion of this study, demonstrated resistance to prior endocrine therapy in the metastatic setting is required; this is defined as:

  * Progressed on prior endocrine therapy in the metastatic setting or,
  * Relapsed on adjuvant endocrine therapy or,
  * Relapsed within 12 months of completing adjuvant endocrine therapy or,
  * If received adjuvant CDK4/6 inhibitor, relapsed at least 2 years after completion of adjuvant CDK4/6 inhibitor
* Washout from prior systemic anti-cancer therapy of at least 3 weeks from chemotherapy or 5 half-lives from oral targeted drugs, and treatment related adverse events recovered to grade 1 (except for alopecia) before the start of study treatment. Washout from prior radiation therapy of at least 2 weeks before the start of the study treatment. Washout from prior endocrine therapy is not required
* Age >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of copanlisib in combination with abemaciclib and fulvestrant in patients < 18 years of age, and because breast cancer is rare in children, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL (no more than 7 days before starting study treatment)
* Absolute neutrophil count >= 1,500/mcL (no more than 7 days before starting study treatment)
* Platelets >= 100,000/mcL (no more than 7 days before starting study treatment)
* Hemoglobin >= 8.0 g/dL (no more than 7 days before starting study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (=< 3 x institutional upper limit of normal for patients with Gilbert syndrome) (no more than 7 days before starting study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal (=< 5 x institutional upper limit of normal for patients with liver involvement) (no more than 7 days before starting study treatment)
* Glomerular filtration rate >= 30 mL/min according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula (no more than 7 days before starting study treatment)
* Lipase =< 1.5 x upper limit of normal (ULN) (no more than 7 days before starting study treatment)
* International normalized rate (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN (except those on anti-coagulation therapy) (no more than 7 days before starting study treatment)
* Hemoglobin (Hb)A1c =< 8.5% or fasting glucose =< 120 mg/dL on at least 2 occasions within 14 days prior to registration if diabetic (no more than 7 days before starting study treatment)
* Left ventricular ejection fraction (LVEF) >= 50%
* Patients may be postmenopausal or premenopausal women on or planned to receive gonadotropin-releasing hormone (GnRH) agonist
* The effects of copanlisib on the developing human fetus are unknown. For this reason and because maternal toxicity, developmental toxicity and teratogenic effects have been observed in nonclinical studies and PI3K inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after the last dose of copanlisib. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of copanlisib administration
* Ability to understand and willing to sign a written informed consent document (or legally authorized representative, if applicable). Patient must agree to research team access to prior breast cancer diagnosis and treatment records, as well as reports of clinical tumor and blood sequencing results
* Patients with a history of treated brain metastases are allowed in the phase I portion of the trial provided there is no disease progression symptomatically and by imaging within 28 days prior to registration AND if the patient is off steroids
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

Exclusion Criteria:

* For patients enrolling to the randomized phase 2 portion of the study, prior treatment with a CDK4/6 inhibitor or fulvestrant, or a PI3K inhibitor in the metastatic setting is not allowed
* Patients who have had chemotherapy within 3 weeks or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who are receiving any other investigational agents
* Immunosuppressive therapy is not allowed while on study
* Receiving anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to copanlisib, PI3K inhibitors, or other agents used in study
* For the randomized phase 2 portion of the study, patients with brain metastasis or a history of brain metastasis are not eligible

  * For the phase 1 portion of the study, patients with progressive brain metastases should be excluded because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs)
* Copanlisib is primarily metabolized by CYP3A4. Therefore, the concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, St. John's wort) are not permitted from 14 days prior to enrollment until the end of the study

  * It is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not permitted while on study. Previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days prior to the computed tomography (CT)/magnetic resonance imaging (MRI) screening. If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose before the screening. Patients may be using topical or inhaled corticosteroids. Short-term (up to 7 days) systemic corticosteroids above 15 mg prednisolone or equivalent will be allowed for the management of acute conditions (e.g., treatment non-infectious pneumonitis)
* Major surgical procedure or significant traumatic injury (as judged by the investigator) within 28 days before start of treatment, or have not recovered from major side effects, open biopsy within 7 days before start of treatment
* Uncontrolled intercurrent illness, including but not limited to, symptomatic congestive heart failure (> New York Heart Association [NYHA] class 2), unstable angina pectoris, new-onset angina, uncontrolled hypertension despite optimal medical management, seizure disorder requiring medication, or psychiatric illness/social situations that would limit compliance with study requirements
* Myocardial infarction < 6 months before start of treatment
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* Proteinuria >= grade 3 as assessed by a 24-hour (h) protein quantification or estimated by urine protein: creatinine ratio > 3.5 on a random urine sample
* History of bleeding diathesis. Any hemorrhage or bleeding event >= grade 3 within 4 weeks prior to the start of study medication
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function
* History of having received an allogeneic bone marrow or organ transplant
* Patients with non-healing wound, ulcer, or bone fracture not due to breast cancer
* Patients with active, clinically serious infections > grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0)
* Patients with HbA1c > 8.5% at screening
* Concurrent diagnosis of pheochromocytoma
* Has undergone blood or platelet transfusion < 7 days prior to start of treatment
* Pregnant women are excluded from this study because copanlisib is a PI3K inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with copanlisib, breastfeeding should be discontinued if the mother is treated with copanlisib. These potential risks may also apply to other agents used in this study
* Hepatitis B (HBV) or hepatitis C (HCV). All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus lab panel. Patients positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) will be eligible if they are negative for HBV DNA, these patients should receive prophylactic antiviral therapy. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV RNA
* HIV positive patients on combination antiretroviral agents that are strong CYP3A4 inhibitors or inducers and who are unwilling or unable to change to antiretroviral therapies without such interactions are ineligible because of the potential for pharmacokinetic interactions with copanlisib, abemaciclib, and fulvestrant. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with history of, or current autoimmune disease are not eligible
* History of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2026-08-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia X Ma, Principal Investigator — Yale University Cancer Center LAO
Locations (14):
- United States (14):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Bellevue Hospital Center, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant): Patients receive 45 mg copanlisib hydrochloride IV over 1 hour on days 1 and 15 and 100 mg abemaciclib PO BID on days 2-28 of cycle 1 and on days 1-28 of subsequent cycles. Patients also receive 500 mg fulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.
- Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant): Patients receive 45 mg copanlisib hydrochloride IV over 1 hour on days 1, 8, and 15 and 150 mg abemaciclib PO twice daily BID for 5 days each week (2 days off). Patients also receive f500 mg ulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.
- Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant): Patients receive 45 mg copanlisib hydrochloride IV over 1 hour on days 1 and 15 and 100 mg abemaciclib PO twice daily BID for 5 days each week (2 days off). Patients also receive 500 fulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.
- Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant): Patients receive 45 mg copanlisib hydrochloride IV over 1 hour on days 1, 8, and 15 and 100 mg abemaciclib PO twice daily BID for 5 days each week (2 days off). Patients also receive 500 mg fulvestrant IM on days 2 and 16 of cycle 1, and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo an ECHO or MUGA scan during screening. Patients also undergo blood sample collection pre-treatment, cycle 1 days 1, 8, 15, and 22, cycle 2 day 1, cycle 4 day 1, cycle 7 day 1, and then every 3 cycles thereafter and at time of progression. Patients undergo tissue biopsy pre-treatment and optionally on cycle 1 day 15 and at the time of progression. Patients also undergo imaging at screening and at the completion of cycle 3, then every 3 cycles thereafter.
Period: Overall Study
Arm/Group | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant)
Started | 7 | 3 | 7 | 7
Completed | 7 | 3 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were not any subjects enrolled in the Phase II portion of the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant) | Total
Number analyzed (Participants) | 7 | 3 | 7 | 7 | 24
Age, Continuous [Median (Full Range); unit: years] | 58 [44 to 68] | 62 [59 to 69] | 56 [40 to 68] | 63 [42 to 78] | 59 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 7 | 7 | 23
  Male | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 3 | 7 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 7 | 2 | 5 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 7 | 7 | 24

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity (DLT)
Description: DLT will be determined based on the incidence, intensity and duration of adverse events (AEs) that are related to the drug combinations and occur within 28 days of drug administration. The severity of AEs will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. AEs will be summarized by counts and percentages, overall as well as by dose levels and by patient characteristics.
Time Frame: Up to 28 days from drug administration
Population: 1 subject in Phase I Part A Dose Level 1 was not evaluable due to copanlisib not being held per protocol. 1 subject in Phase I Part B Dose Level 1b and 1 subject in Phase I Part B Dose Level 2b were not evaluable as they had cycle 1 dosing errors.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant)
Number analyzed (Participants) | 6 | 3 | 6 | 6
Participants | 1 | 2 | 1 | 2

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Radiographic disease recurrence/progression will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Will be estimated by the Kaplan-Meier (KM) product limit method and survival difference will be compared between the two arms by stratified log rank test. Hazard ratio with 95% confidence interval (CI) will be estimated between the two arms from the stratified Cox proportional hazard model, without and with adjustment for patient characteristics.
Time Frame: Time from randomization to the event of disease recurrence/progression or death due to any cause, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant)
Number analyzed (Participants) | 7 | 3 | 7 | 7
months | 5.9 [2.5 to 14.8] | 7.9 [2.3 to NA] — Due to an insufficient number of participants who have progressed (events), the upper CI bound is not estimable. | 19.3 [2.8 to NA] — Due to an insufficient number of participants who have progressed (events), the upper CI bound is not estimable. | 18.7 [1.8 to NA] — Due to an insufficient number of participants who have progressed (events), the upper CI bound is not estimable.
Statistical Analysis 1: Comparison: Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) vs Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) vs Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) vs Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant); Test type: Other — This test is used to compare the survival distributions of different groups in a survival analysis. It's a nonparametric test; p = 0.5060, Log Rank

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Will be defined as the proportion of response-evaluable patients who achieve complete response (CR) or partial response (PR) and assessed by RECIST 1.1 criteria. Will be estimated with a 95% exact CI and difference between the two arms will be compared by Fisher's exact test. Raw and adjusted odds ratio (OR) will be derived with 95% CI from logistic regression without and with adjustment for patient characteristics.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant)
Number analyzed (Participants) | 7 | 3 | 7 | 7
Participants | 1 | 0 | 2 | 2

4. Secondary Outcome: Clinical Benefit Rate
Description: Will be defined as the proportion of response-evaluable patients who achieve CR or PR or stable disease (SD) for at least 6 months and assessed by RECIST 1.1 criteria. Will be estimated with a 95% exact CI and difference between the two arms will be compared by Fisher's exact test. Raw and adjusted OR will be derived with 95% CI from logistic regression without and with adjustment for patient characteristics
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Part A Dose 1 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part A Dose 2 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose 1b (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose 2b (Copanlisib, Abemaciclib, Fulvestrant)
Number analyzed (Participants) | 7 | 3 | 7 | 7
Participants | 3 | 0 | 3 | 2

5. Secondary Outcome: Overall Survival
Description: Will be assessed by RECIST 1.1 criteria. Will be estimated by the KM product limit method and survival difference will be compared between the two arms by stratified log rank test. Hazard ratio with 95% CI will be estimated between the two arms from the stratified Cox proportional hazard model, without and with adjustment for patient characteristics.
Time Frame: Time of randomization to time of death due to any cause or latest follow-up, whichever earlier, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant)
Number analyzed (Participants) | 7 | 3 | 7 | 7
months | 14.8 [2.5 to NA] — Due to an insufficient number of participants who have experienced death (events), the upper CI bound is not estimable. | 12.2 [2.3 to NA] — Due to an insufficient number of participants who have experienced death (events), the upper CI bound is not estimable. | NA [20.1 to NA] — Due to an insufficient number of participants who have experienced death (events), the median and upper CI bound is not estimable. | NA [3.6 to NA] — Due to an insufficient number of participants who have experienced death (events), the median and upper CI bound is not estimable.
Statistical Analysis 1: Comparison: Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) vs Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) vs Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) vs Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2989, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from start of treatment through the end of treatment visit. Patients removed due to unacceptable AE(s), were followed until resolution or stabilization of the AE. Median AE length of follow-up was 126 days (full range 28-710 days). All-cause mortality was collected from start of treatment to death due to any cause or latest follow-up, whichever earlier. Overall median length of follow-up was 439 days (full range 66-1198 days).
Arm/Group | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant)
All-Cause Mortality (participants affected / at risk) | 5/7 | 3/3 | 2/7 | 2/7
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/3 | 4/7 | 5/7
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) (N=7) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) (N=3) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) (N=7) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant) (N=7)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Adult respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chest wall necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Part A Dose Level 1 (Copanlisib, Abemaciclib, Fulvestrant) (N=7) | Phase I Part A Dose Level 2 (Copanlisib, Abemaciclib, Fulvestrant) (N=3) | Phase I Part B Dose Level 1b (Copanlisib, Abemaciclib, Fulvestrant) (N=7) | Phase I Part B Dose Level 2b (Copanlisib, Abemaciclib, Fulvestrant) (N=7)
Anemia (Blood and lymphatic system disorders) | 7 | 1 | 4 | 6
Blood Lymph - other - macrocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac disorders - Other - Brain Natriuretic Peptide Increased (Cardiac disorders) | 0 | 0 | 0 | 1
First-degree atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 3
Ear and Labyrinth - Other - Ear Drainage (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Floaters (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 3 | 5 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 1 | 0
GI disorders - Other - Hematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Investigations - Other, specify - Loose Stool (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 1 | 5
Nausea (Gastrointestinal disorders) | 6 | 3 | 5 | 5
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2 | 3
Chills (General disorders) | 0 | 0 | 0 | 1
Edema limbs (General disorders) | 1 | 1 | 2 | 2
Edema trunk (General disorders) | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 5 | 3 | 4 | 7
Fever (General disorders) | 1 | 1 | 2 | 4
Flu-like symptoms (General disorders) | 1 | 0 | 0 | 0
Generalized edema (General disorders) | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Pain (General disorders) | 3 | 1 | 2 | 0
Fungemia (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex reactivation (Infections and infestations) | 1 | 0 | 0 | 1
Infections & infestations - Other - Pseudomonas Aeruginosa (Infections and infestations) | 0 | 1 | 0 | 0
Infections & infestations - Other - Viral Illness (Infections and infestations) | 0 | 0 | 2 | 0
Infections and Infestations other Covid-19 Infection (Infections and infestations) | 0 | 0 | 1 | 3
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ALT increased (Investigations) | 6 | 1 | 4 | 3
AST increased (Investigations) | 4 | 1 | 4 | 1
Alkaline phosphatase increased (Investigations) | 4 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 1
Cardiac troponin T increased (Investigations) | 0 | 0 | 0 | 2
Creatinine increased (Investigations) | 2 | 1 | 3 | 5
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1
Elevated lactate dehydrogenase (Investigations) | 0 | 0 | 0 | 1
Investigations - Other, specify - Ionized Calcium Decreased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 6 | 0 | 2 | 5
Neutrophil count decreased (Investigations) | 5 | 0 | 4 | 3
Platelet count decreased (Investigations) | 4 | 1 | 2 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 1
Weight loss (Investigations) | 2 | 0 | 1 | 2
White blood cell decreased (Investigations) | 6 | 1 | 3 | 6
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Metabolism and nutrition - Other - Non-Onion Gap Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal/connect tissue -Other - Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal/connect tissue -Other - Pain In Sacrum (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal/connect tissue -Other - Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 3 | 0 | 2 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal & urinary disorders - Other - Bun Increase (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal & urinary disorders - Other - Tingling Sensation Of Bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 3
Skin & subcutaneous tissue -Other - Desquamation Of Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin & subcutaneous tissue -Other - Erythematous Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 0 | 4 | 6
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03939897/Prot_SAP_001.pdf
  • Informed Consent Form: Research Study Informed Consent Document-Phase 1 (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03939897/ICF_002.pdf
  • Informed Consent Form: Research Study Informed Consent Document-Phase 2 (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03939897/ICF_003.pdf